CLINICAL TRIAL: NCT06736379
Title: Study of Intratumoral Injections of VLPONC-01 in Head and Neck Cancer
Brief Title: Intratumoral Delivery of Viral Replicon (saRNA) Particles Expressing IL-12 in Head and Neck Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VLP Therapeutics (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VLPONC-01; SYNERNA-01 (Other: VLP Therapeutics, Inc.)
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancers- Squamous Cell; Head and Neck Cancer; Solid Tumors; HNSCC; SCC - Squamous Cell Carcinoma; SCCHN; Head Neck Cancer; Head and Neck Squamous Cell Cancer; Squamous Cell Carcinoma of the Head and Neck; Squamous Cell Carcinoma, Head And Neck; Squamous Cell Head and Neck Carcinoma; Oral Cavity; Oral Cavity Carcinoma
Keywords: Virus-like particle; VLP; IL-12; Interleukin 12; Intratumoral; VRP; Viral Replicon Particle; saRNA; VRP-encapsulated; IT injection; pembrolizumab; anti-PD-1; tumor resection surgery; tumor resection; Self-amplifying RNA; Multiple inoculations directly into the tumor; Keytruda; viral particles per injection; viral particles; macrophage
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell; Mouth Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Dose de-escalation Model
Masking Description: Cohort A is nonrandomized. Cohort C subjects will be randomized into 3 different treatment groups. Both investigator and subject will not be blinded to treatment group assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (1 x 10^9 viral particles per injection) (Experimental): Recurrent or Metastatic Head and Neck Cancer not scheduled for tumor resection surgery, 4 doses VLPONC-01 administered IT once weekly, with an additional follow-up safety visit 30 and 90 days post the final injection.
  Interventions: Biological: VRP-encapsulated saRNA encoding IL-12 (1 x 10^9 viral particles per injection)
- Cohort C - Group 1 (1 x 10^9 viral particles per injection plus Pembrolizumab) (Experimental): Head and Neck Squamous Cell Carcinoma Patients scheduled for tumor resection surgery, 4 doses VLPONC-01 administered IT once weekly and 2 doses of 200mg neoadjuvant Pembrolizumab IV 3 weeks apart prior to tumor resection surgery, follow-up safety visit 30 days post-surgery and 90 days post final treatment.
  Interventions: Biological: VRP-encapsulated saRNA encoding IL-12 (1 x 10^9 viral particles per injection); Drug: Pembrolizumab (KEYTRUDA®)
- Cohort C - Group 2 (3 x 10^8 viral particles per injection plus Pembrolizumab) (Experimental): Head and Neck Squamous Cell Carcinoma Patients scheduled for tumor resection surgery, 4 doses VLPONC-01 administered IT once weekly and 2 doses of 200mg neoadjuvant Pembrolizumab IV 3 weeks apart prior to tumor resection surgery follow-up safety visit 30 days post-surgery and 90 days post final treatment.
  Interventions: Drug: Pembrolizumab (KEYTRUDA®); Biological: VRP-encapsulated saRNA encoding IL-12 (3 x 10^8 viral particles per injection)
- Cohort C - Pembrolizumab only (Experimental): Head and Neck Squamous Cell Carcinoma Patients scheduled for tumor resection surgery, 2 doses of 200mg neoadjuvant Pembrolizumab IV 3 weeks apart prior to tumor resection surgery, follow-up safety visit 30 days post-surgery and 90 days post final treatment.
  Interventions: Drug: Pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Biological: VRP-encapsulated saRNA encoding IL-12 (1 x 10^9 viral particles per injection) — Weekly IT injections of 1 x 10^9 viral particles of VLPONC-01
  Other Names: VLPONC-01; IL-12 saRNA; VRP-IL-12
  Arms: Cohort A (1 x 10^9 viral particles per injection); Cohort C - Group 1 (1 x 10^9 viral particles per injection plus Pembrolizumab)
Drug: Pembrolizumab (KEYTRUDA®) — 200mg twice 3 weeks apart IV
  Other Names: Pembrolizumab
  Arms: Cohort C - Group 1 (1 x 10^9 viral particles per injection plus Pembrolizumab); Cohort C - Group 2 (3 x 10^8 viral particles per injection plus Pembrolizumab); Cohort C - Pembrolizumab only
Biological: VRP-encapsulated saRNA encoding IL-12 (3 x 10^8 viral particles per injection) — Weekly IT injections of 3 x 10^8 viral particles of VLPONC-01
  Other Names: VLPONC-01; VRP-IL-12; IL-12 saRNA
  Arms: Cohort C - Group 2 (3 x 10^8 viral particles per injection plus Pembrolizumab)

SUMMARY:
The goal of this clinical trial is to assess the safety and tolerability of a virus replicon particle (VRP) encapsulated saRNA encoding IL-12 when injected into in head and neck cancer patients. The main questions being addressed are:

The safety and tolerability of intratumoral (IT) injections of VRP-encapsulated saRNA encoding IL-12 (VLPONC-01)

The tumor response to IT injections of VLPONC-01

The tumor response due to the combination of IT injections of VLPONC-01 and system IV administration of neoadjuvant pembrolizumab (anti-PD-1) treatment

Researchers will compare neoadjuvant pembrolizumab alone to the combination therapy to see if the combination enhances tumor responses.

DETAILED DESCRIPTION:
The study is an Open label, Phase I study to determine the safety of IT injected VLPONC-01 as a therapeutic agent in subjects with non-resectable and resectable Head and Neck Cancer Squamous Cell Carcinomas (HCSCC), and secondarily to assess pathologic response and radiological response (assessed by RECIST 1.1 criteria) in the primary tumor and regional lymph nodes. Researchers also will explore tumor microenvironment changes in cytokine levels and cellular responses.

There will be three distinct cohorts enrolling sequentially:

Cohort A: Researchers will enroll unresectable or recurrent/metastatic head and neck cancer with at least 1 injectable tumor not scheduled for tumor resection surgery who will receive four doses of VLPONC-01.

Cohort C: Researchers will enroll HCSCC patients scheduled for tumor resection surgery who will receive four doses of VLPONC-1 and two doses of neoadjuvant pembrolizumab or only two doses of neoadjuvant pembrolizumab prior to tumor resection surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort A - Unresectable or recurrent/metastatic head and neck cancer with at least 1 injectable tumor not scheduled for tumor resection surgery. With one the following prior treatments:

   Subjects must have received a platinum containing chemotherapy regimen, 5-Fluorouracil chemotherapy, taxane based chemotherapy, cetuximab or gemcitabine for treatment of primary tumor in locally advanced, or metastatic settings.

   Subjects must have received an anti-PD-1/ PD-L1 as monotherapy or in combination with chemotherapy.

   Subjects must have progressed following therapy with at least one PD-1 or PD-L1 checkpoint inhibitor (regardless of PD-L1 expression status).

   Prior progression on a PD-1 or PD-L1 checkpoint inhibitor should be unequivocal; progression that occurs within the first 8 weeks of treatment on these agents should be confirmed with a second CT at least 4 weeks apart (to exclude pseudo-progression).

   Patients with activating EGFR mutation or ALK rearrangement which is expected to be responsive to available tyrosine kinase inhibitor therapy, therefore these subjects must have been previously treated with an applicable tyrosine kinase inhibitor.

   OR Cohort C - Patients with at least 1 measurable resectable lesion clinical stage I-IVb (cT1-4, N0-3) (AJCC, 8th Edition) (Amin, 2017), Histologically or cytologically confirmed HNSCC. Scheduled to undergo tumor surgical resection of the primary tumor.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-1, and adequate bone marrow and organ function.
3. Primary tumors should be amenable to intratumoral (IT) injection >1 cm diameter. This will be determined by the Protocol Director, or the surgeon involved.
4. Subjects with either a local recurrence or a new primary tumor will be allowed.
5. Age ≥ 18 years.
6. Have acceptable organ and marrow function defined as follows:

   Absolute neutrophil count ≥ 1,500/mcL Platelets ≥ 100,000/mcL Hemoglobin ≥ 8.0 g/dL (Note: use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dL is acceptable) Total bilirubin ≤2x institutional upper limit of normal (ULN) AST(SGOT) or ALT(SGPT) ≤ 3.0x institutional ULN
7. Ability to understand and the willingness to provide written informed consent.
8. Life expectancy > 12 weeks (about 3 months).
9. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Tumors which are not feasible for injections include high risk lesions that are near vital organs or important neurovascular structures, as determined by the Protocol Director or involved surgeon.
2. Women of childbearing potential must have a negative serum β-hCG pregnancy test within 7 days prior to the administration of the first study treatment and/or urine pregnancy 48 hours prior to the administration of the first study treatment. Both sexually active women of childbearing potential and males (and their female partners) patients must agree to use two methods of effective contraception, one of them being a barrier method, or to abstain from sexual activity during the study and for at least 6 months after last dose of study drugs.
3. Patients expected to receive other anti-cancer medication such as, chemotherapy, immunotherapy, biologic therapy, targeted therapy, monoclonal antibodies, hormonal therapy (other than leuprolide or other GnRH agonists) prior to surgery and where all acute toxicity of prior treatments have not resolved.
4. Participation in another clinical study with an investigational product during the last 30 days.
5. Uncontrolled intercurrent illness including, that do not respond to active medical intervention.
6. Current or prior use of immunosuppressive medication within 28 days before the first dose of injection, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone or an equivalent corticosteroid.
7. If applicable: Women who are breastfeeding.
8. History of allogenic organ transplant that requires use of immunosuppressives.
9. Subject has active or uncontrolled infection including known HIV infection or known chronic hepatitis B or C.
10. Any condition that, in the investigator's opinion, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
11. Uncontrolled intercurrent illness including those that do not respond to active medical intervention.
12. Any contraindication to the use of known history of hypersensitivity to any immune therapy's drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | First injection to 90-day follow-up visit post-final injection (Cohort A) or post-surgery (Cohort B and Cohort C)
  To assess the safety and tolerability of VLPONC-01. Safety will be based on the occurrence of any grade 3 or higher drug-related adverse events from the VLPONC-01 injections for non-surgery patients and any grade 3 or higher drug-related adverse events that result in a delay to tumor resection surgery.

SECONDARY OUTCOMES:
Levels of circulating IL-12 | First injection to 30-day follow-up visit post-final injection (Cohort A) or post-surgery (Cohort B and Cohort C)
  To assess the circulating blood levels of IL-12 after VLPONC-01 treatment compared to baseline to determine the occurrence and safety profile of potential systemic inflammatory responses.
VLPONC-01 levels in tumor tissue | First injection to tumor resection surgery
  To detect levels of VLPONC-01 RNA in surgically resected tissue.
Tumor response | First injection to tumor resection surgery
  To assess the primary tumor response by radiological imaging and pathological analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Fred M Baik, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No